CLINICAL TRIAL: NCT06204991
Title: Phase 1 Study to Evaluate the Safety and Efficacy of TILs Transduced With IL-7 (ADP-TILIL7) in Patients With Locally Advanced or Metastatic Melanoma
Brief Title: To Evaluate the Safety and Efficacy of ADP-TILIL7 in Patients With Locally Advanced or Metastatic Melanoma
Acronym: ADP-TILIL7
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Collaborators: Adaptimmune (Industry)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Professor, M.D., Ph.D., Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM2319
Record Dates: First submitted 2023-12-15; First posted 2024-01-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Melanoma Stage III; Melanoma Stage IV; Melanoma
Keywords: adoptive cell therapy; immunetherapy; genemodified tumor infiltrating lymphocytes; IL-7
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine phosphate; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor-infiltrating lymphocytes genemodified with IL-7 gene for IL-7 production upon Ag engagement (Experimental): Tumor-infiltrating lymphocytes grown ex-vivo from resected tumor tissue and reapplied to the patient via an intravenous infusion.
  Drug: Cyclophosphamide: 2 doses (69 mg/kg) prior to infusion Drug: Fludarabinephosphat 5 doses (25 mg/m2, max. 50 mg) prior to infusion Drug: Proleukin 600.000 IU/kg/dose IL-2 a maximum of 6 doses
  Interventions: Biological: ADP-TILIL7; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Drug: Proleukin

INTERVENTIONS:
Biological: ADP-TILIL7 — Autologous tumor infiltrating lymphocytes genemodified (by a lentiviral vector) to produce IL-7 upon antigen engagement
Drug: Cyclophosphamide — Lymphodepleting Chemotherapy
Drug: Fludarabine Phosphate — Lymphodepleting Chemotherapy
Drug: Proleukin — IL-2

SUMMARY:
The primary objective of this Phase 1 clinical trial is to evaluate the feasibility and tolerability of a novel generation of gene-modified tumor infiltrating lymphocytes (TILs) in a cohort of 10 patients aged 18-75 diagnosed with unresectable or metastatic melanoma. TILs will undergo transduction with the Interleukin-7 (IL-7) gene, for IL-7 production upon antigen engagement.

Participants will undergo:

* screening
* tumor operation following autologous TIL production (incl. transduction) - takes approximately 4-6 weeks
* admission for lymphodepleting chemotherapy (Cyclophosphamide and Fludarabine phosphate), TIL infusion and high-dose IL-2 infusions for a maximum of 6 doses
* Following treatment, patients will undergo systematic and regularly planned assessments, encompassing clinical evaluation, biochemistry analyses, and PET/CT scans. This thorough follow-up regimen will be continued until any of the following events occur: progressive disease, withdrawal from study, or end of study, which spans a duration of 15 years for trials involving genetically modified organisms.

DETAILED DESCRIPTION:
Synopsis:

Over the last decade treatment for malignant melanoma (MM) has seen remarkable progress particularly with checkpoint inhibitors (anti-PD-1 and anti-CTLA-4). The combination of these inhibitors has elevated the 5-year overall survival (OS) from 5 % to 50 %. However, many patients still lack a durable response.

Results from a Phase III trial, conducted in part at CCIT-DK, have illuminated the promising potential of adoptive cell therapy utilizing tumor infiltrating lymphocytes (TILs) in the treatment of malignant melnaoma. In this trial, 168 patients were randomly assigned to receive either standard anti-CTLA-4 treatment or TILs. The outcomes revealed a notably superior overall response rate (ORR) and a higher number of complete responses (CR) among those treated with TILs.

In this phase I study the investigators intend to treat 10 subjects with locally advanced or metastatic MM. Included subjects undergo surgical removal of tumor tissue for TIL manufacturing. During TIL manufacture, the investigators will genetically modify the TILs, and enable them to produce Interleukin-7 (IL-7). This modification is anticipated to confer additional functionality to the TILs enhancing their proliferation and persistence. The lentiviral vector used to integrate the IL-7 gene to the TILs is manufactured and provided by the British/American biotechnological company, Adaptimmune. The genetically modified TILs are therefore called ADP-TILIL7.

Lymphodepleting (LD) chemotherapy is administered 7 days prior to ADP-TILIL7 infusion. ADP-TILIL7 infusion is followed by high dose (HD) Interleukin (IL-2) for a maximum of 6 doses or until tolerance.

Purpose:

The primary objective of this study is to evaluate the tolerability and safety of treatment with ADP-TILIL7. The secondary objective is to assess the clinical effect of the treatment by use of the objective response rate (using RECIST 1.1). Overall survival (OS), progression-free survival (PFS), duration of response (DoR) and disease control rate (DCR) will be determined. In addition to this replication competent lentivirus (RCL) will be monitored.

Exploratory objectives are to characterize the tumor and tumor microenvironment pre- and post infusion, ex by genomic profiling of tumor tissue to investigate the mutational landscape. Furthermore, the expression of tumor-associated immunerelated markers, including markers of phenotype and frequency of tumor infiltrating blood-derived cells. The investigators want to characterize subjects' peripheral blood which includes, but is not limited to, the phenotype and funcitionality of transduced TILs and non-transduced TILs, as well as the pharmacodynamic changes in whole blood and serum pre- and post infusion, which might include gene expression, TCR/B-cell receptor repertoire, cytokines and soluble markers. All this the investigators want to explore to understand factors that can influence response or resistance to ADP-TILIL7 therapy.

Study design:

This is a phase I, First-in-human, study. Ten (10) subjects with locally advanced or metastatic MM will be included and treated at the Department of Oncology, Herlev Hospital. Subjects can be referred from other oncology centers.

Subjects will undergo a comprehensive screening process to confirm subjects' eligibility before enrollment. Included subjects will undergo surgical tumor removal for the subsequent manufacturing of TIL's. TheTIL manifacturing process is expected to take approximately 4-6 weeks. During TIL manufacture, a subset of the TILs will be transduced with genetic material encoding the production of IL-7.

Lymphodepleting chemotherapy, Cyclophosphamide and Fludarabine phosphate, will be administered for 7 days prior to ADP-TILIL7 infusion. ADP-TILIL7 infusion is followed by high-dose IL-2 for a maximum of 6 doses or until tolerance. After the end of treatment, the subjects will be followed with clinical- and imaging controls for up to 15 years.

The inclusion period is set to commence in early 2024, with the goal of enrolling all ten patients within a span of three years. The study's completion is defined as the moment when the last subject reaches and complete the 12 months follow-up visit. The study ends once all treated subjects complete 15 years of follow-up, passes away or withdraw from the study.

The study will be monitored by the Good Clinical Practice (GCP)-unit of the Capital Region of Denmark. The Danish Medicines Agency, The GCP-unit, and Adaptimmune are allowed to audit this trial.

Population:

This study targets subjects aged 18 to 75, histologically confirmed with malignant melanoma who have experienced progression following at least one line of immune checkpoint inhibitor in the advanced or metastatic setting. Eligibility is contigent on meeting specific inclusion criteria, including acceptable performance status, kidney- and liver function, and the absence of major co-morbidities. Crucially, treatment will proceed only for the subjects with successful manufacturing of TILs. Previous clinical trials have demonstrated a success rate of TIL manufacturing from malignant melanoma exceeding 90%.

Toxicity:

The amount of toxicity caused by ADP-TILIL7 is not known. The systemic treatment with IL-7 infusion has been used in treatment of several malignancies and HIV and as an adjunct to allogeneic stem cell transplantation. In these studies, IL-7 has exhibited a generally well-tolerated safety profile. At CCIT-DK investigators boast substantial experience in treating subjects with TILs that have not been genetically modified. TIL therapy has generally been well-tolerated, with most adverse events expected to be associated with chemotherapy and high-dose IL-2 treatment.

Dosing in the first three subjects will be staggered. Each subject will have safely completed a minimum observation period of 14 days from the ADP-TILIL7 infusion before lymphodepletion of the next subject commences.

Toxicity assessment, including evaluation of treatment limiting toxicity (TLTs), will be performed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The TLT observation period will be during the first 21 days following the ADP-TILIL7 infusion.

Evaluation of clinical response:

Subjects enrolled in the study will undergo comprehensive clinical evaluations during treatment and hospitalization as well as 6, 12 and 24 weeks post-treatment with ADP-TILIL7. Thereafter clinical evaluation will take place every 3 months the first two years (year 1-2), every 6 months year 3-5, followed by evaluations every 12 months year 6-15. Diagnostic imaging, preferably PET/CT scans, will be conducted before the treatment initiation, and in conjunction with the clinical evaluations, commencing 6 weeks post-TIL treatment.

Immunological response evaluation:

Blood samples for research purposes will be systematically collected at Baseline, pre- and post-TIL infusion (day 0), during IL-2 (up to a maximum 3 days), before discharge and at week 6, week 12 and the final collection 12 months post-ADP-TILIL7/progressive disease/withdrawal whichever occurs first. Blood samples for research purposes will be selectively collected, contigent upon feasibility as assessed by the investigator. Biopsies from metastatic tumor tissue will be systematically obtined at key time points: before treatment initiation, 6 weeks post-treatment and, if applicable and deemed safe, in case of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* All the criteria listed in the following need to be met before patient inclusion.

  1. Histologically confirmed inoperable or metastatic melanoma (stage IIIc or IV).
  2. Progressive disease after standard treatment with PD-1 check-point inhibition or combination of aforementioned with CTLA-4 check-point inhibition.
  3. Age: 18 - 75 years at time of signed Informed consent.
  4. ECOG performance status of ≤ 1 (Appendix 2).
  5. Is fit for tumor resection and has at least one lesion (> 1 cm3) available for surgical resection for manufacture of TIL.
  6. At least one measurable parameter in accordance with RECIST 1.1 -criteria (excluding lesion to be resected).
  7. LVEF assessment with documented LVEF ≥50% by either TTE (transthoracic echocardiography) or MUGA (multigated acquisition scan).
  8. Sufficient organ function, including:

     * Absolute neutrophil count (ANC) ≥ 1.500 /µl
     * Leucocyte count ≥ lower normal limit
     * Platelets ≥ 100.000 /µl and <700.000 /µl
     * Hemoglobin ≥ 6.0 mmol/l
     * eGFR > 70 ml/min*
     * S-bilirubin ≤ 1.5 times upper normal limit (Exception: Subjects with liver metastasis ≤ 2.5 × ULN)
     * ASAT/ALAT ≤ 2.5 times upper normal limit (Exception: Subjects with liver metastasis ≤ 5.0 × ULN)
     * Alkaline phosphatase ≤ 5 times upper normal limit
     * Lactate dehydrogenase ≤ 5 times upper normal limit
     * Sufficient coagulation: APPT<40 and INR<1.5
* * In selected cases it can be decided to include a patient with an eGFR < 70 ml/min with the use of a reduced dose of chemotherapy.

  9. Signed statement of consent after receiving oral and written study information 10. Willingness to participate in the planned controls and capable of handling toxicities.

  11. Subject must receive T-cell therapy as the next therapy following tumor resection, unless bridging therapy is administered:
  * Bridging therapy is discouraged. However, if in the opinion of the Investigator, the subject requires immediate therapy after tumor resection, the subject may receive bridging therapy for the period during which the subject is awaiting the manufacture of TIL-infusion product. Bridging therapy may be a continuation of the therapy the subject was receiving prior to tumor resection or may be a new therapy.
  * Following this bridging therapy, the subject must adhere to the mandatory washout periods (exclusion criterion 1) and must continue to have measurable disease prior to receiving T-cell therapy.

    12. Age and Reproductive Status:
  * Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test AND must agree to use an effective method of contraception starting at the first dose of chemotherapy for at least 12 months. WOCBP must also agree to refrain from egg donation, storage, or banking during these same time periods. The following are considered safe methods of contraception:
* Hormonal anticonception (birth control pills, spiral, depot injection with gestagen, subdermal implantation, hormonal vaginal ring and transdermal depot patch)
* Intrauterine device
* Surgical sterilization
* Surgical sterilization of male partner with verification of no sperm after the procedure
* Menopause (for more than 12 months) o Male subjects must be surgically sterile or agree to use a double-barrier contraception method or abstain from sexual activity with an WOCBP starting at the first dose of chemotherapy and for 6 months thereafter. Male subjects must also agree to refrain from sperm donation, storage, or banking.

Exclusion Criteria:

* Patients will be excluded if they meet one of the criteria's listed below

  1. Subject has received or plans to receive the following therapy/treatment prior to tumor resection (TR) or lymphodepleting chemotherapy (LDC):

     * Cytotoxic chemotherapy: Washout period 3 weeks before TR and LDC
     * Small molecules/TKI: Washout period 1 week before TR and LDC
     * Immune therapy (monoclonal AB therapy, CPI and biologics): 2 weeks before TR and LDC
     * Prior T-cell therapy, including gene therapy using an integrating vector
     * Corticosteroids at dose equivalent > 10 mg prednisone or any other immunosuppressive therapy. 2 weeks before TR and LDC. Note: Use of topical steroids is not an exclusion
     * Investigational treatment: 4 weeks or 5 half-lives, whichever is shorter before TR and LDC
     * Radiation to the pelvis and/or multiple bones containing ≥ 25% of bone marrow: 4 weeks before TR and LDC
     * Whole brain radiotherapy or brain stereotactic radiosurgery: 4 weeks before TR and LDC
     * Radiotherapy to the target lesions: 3 months prior to TIL-infusion. A lesion with unequivocal progression post-radiotherapy may be considered a target lesion.
  2. A history of prior malignancies. Patients treated for another malignancy can participate if they are without signs of disease for a minimum of 2 years after treatment. Subjects with curatively treated ductal carcinoma in situ (DCIS or LCIS) breast cancer for which they are taking hormonal therapy is acceptable. Resectable squamous or basal cell carcinoma of the skin is acceptable.
  3. Patients with metastatic ocular/mucosal or other non-cutaneous melanoma. Unknown primary melanoma is eligible.
  4. Toxicity from previous anti-cancer therapy must have resolved to ≤ Grade 1 or baseline prior to enrollment (except for non-clinically significant toxicities e.g., alopecia, vitiligo).

     Subjects with Grade 2 toxicities who are deemed stable or irreversible (e.g., peripheral neuropathy) can be enrolled.
  5. Patients who have more than 2 CNS metastases or who have any CNS lesion that is symptomatic, greater than 1 cm in diameter or show significant surrounding edema on MRI scan will not be eligible until they have been treated and demonstrated no clincal or radiologic CNS progression for at least 2 months.
  6. The following patients will be excluded because of inability to receive high dose interleukin-2:

     * History of coronary revascularization
     * Patients with clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, 2o or 3o heart block
     * Documented FEV-1 less than or equal to 60% predicted value for patients with: A prolonged history of cigarette smoking (greater than 20 pack years), large tumor burden in the lungs or Symptoms of respiratory distress.
  7. Known hypersensitivity to one of the active drugs or one or more of the excipients.
  8. Severe medical conditions, such as severe asthma/COLD, significant cardiac disease, poorly regulated insulin dependent diabetes mellitus among others.
  9. Acute/chronic infection with HIV, hepatitis, syphilis among others.
  10. Severe allergies or previous anaphylactic reactions.
  11. Active autoimmune or immune-mediated disease that has not yet resolved. Subjects with the following will be eligible:

      * Immune-mediated AEs secondary to immunotherapy which has resolved to ≤ Grade 1 off steroids;
      * Hypothyroidism, Type I diabetes, adrenal insufficiency, or pituitary insufficiency that are stable on replacement therapy;
      * Disorders such as asthma, vitiligo, psoriasis, or atopic dermatitis that are well controlled without requiring systemic immunosuppression;
      * Other stable immune conditions that do not require prednisone higher than 10 mg/day or their equivalent dose for other corticosteroid agents may be acceptable with the agreement of the Sponsor.
  12. Pregnant women and women breastfeeding.
  13. Subject who, in the opinion of the Investigator, will be unlikely to fully comply with protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability of the treatment | Through study completion, an average of 1 year
  Fraction of subjects experiencing grade >/= 3 AE
Feasibility of the treatment | Through study completion, an average of 1 year
  Measured by the number of subjects who undergo surgery and succesfully undergo ADP-TILIL7-infusion

SECONDARY OUTCOMES:
Objective response rate | Until progression up to 15 years
  Defined as the proportion of subjects who have a partial or complete response to therapy. Response evaluation criteria in solid tumors, RECIST 1.1. criterias assesed by CT scan
Overall survival | 15 years
  Time from initiation of treatment to death
Progression free survival | Until progression or death up to 15 years
  Time from initiation of treatment until first evidence of disease progression or death
Duration of response | 15 years
  Time from initiation of treatment to disease progression or death in subjects who achieve complete or partial response
Disease control rate | 15 years
  The percentage of subjects whose therapeutic intervention has led to a complete response, partial response or stable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Prof., M.D., Study Director — Study Director, CCIT-DK, Depth of Oncology, Herlev Hospital; Cecilie D Vestergaard, M.D., Principal Investigator — Clinical research assistant, CCIT-DK, Depth of Oncology, Herlev Hospital
Locations (1):
- Department of Oncology, Herlev, Denmark